CLINICAL TRIAL: NCT07003048
Title: Life vs. Digital Music Interventions Performed by Professionals Throughout Pregnancy to Increase Mental Health for Mothers and Their Offspring
Acronym: MusicMums
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clara Angela Foundation (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Birgit Arabin, MD, PhD, Professor of OBGYN, Head of the Clara Angela Foundation, Clara Angela Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eth-SB-24-086
Record Dates: First submitted 2025-04-05; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Mental Health; Maternal and Child Health Outcomes
Keywords: Music intervention; Pregnancy; Stress; Mental health; Anxiety; Depression; Fetal development
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression | interventions — Singing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live music intervention (Experimental): Singing and dancing in small groups combined with live concerts througout pregnancy
  Interventions: Behavioral: Singing, dancing in small groups and active listening to live music at the Berlin Philharmony building
- Digital music intervention (Active Comparator): Digitalized version of singing and dancing workshops combined with recorded concerts offered to women at home throughout pregnancy
  Interventions: Behavioral: Singing, dancing in small groups and active listening to live music at the Berlin Philharmony building

INTERVENTIONS:
Behavioral: Singing, dancing in small groups and active listening to live music at the Berlin Philharmony building — Pregnant women are invited from 12 gestational weeks onwards to participate in active and passive interventions following a protocol derived from our feasibility study. The following interventions take place:
  LIVE GROUP
  1. concerts customized for pregnant women by professionals. They talk before and in between the concerts about the meaning of the music with the study attendants. The sessions take around one hour.
  2. workshops in singing led by professional coaches performed in small groups within the Philharmonic building involving pregnant women to actively learn melodies of songs which they can repeat at home on a daily basis.
  3. workshops in dancing led by professional coaches performed in small groups within the Philharmonic building involving pregnant women to actively learn to move with music which they can repeat at home on a daily basis.
  DIGITAL GROUP The described interventions are all digitalized with interviews encouraging the second group to participate from home.

SUMMARY:
This prospective study was preceded by an extensive feasibility study between 2021-2024. Thereby, pregnant women were exposed to live music and a variety of creative workshops such as vibration, modelling, creative writing, singing, dancing and active listening to concerts from 12 gestational weeks onwards up to delivery at two-week intervals. The investigators detected significant changes in affection detected by the PANAS-test, cortisol from buccal swabs, and maternal heart rate variability before and after the interventions. Similarly, the investigators could detect significant changes by validated questionnaires for maternal stress (PSS), maternal anxiety detected by STAI and the risk of depression detected by EPDS.

Therefore, from January 2025 onwards, the investigators integrated "only" concerts and workshops in singing and dancing as relevant interventions. In a comparative prospective study, the investigators now want to study, whether the effects of life participation within the Philharmonic building at approximately 2-week intervals would have the same short-term and medium-term effects as in pregnant women following the same digitalized interventions from home (DIGITALIZED versus LIVE INTERVENTION = DL). This would offer the chance to reach pregnant women in regions with high needs for interventions to reduce stress during pregnancy, such as in areas involved in wars, environmental disasters or other stressful life conditions.

The primary outcomes are short-term differences in affection measured immediately before and after all interventions, and differences in cortisol from buccal swabs, measured twice after concerts during pregnancy.

The secondary outcomes are the medium-term changes throughout pregnancy in validated questionnaires of PSS, STAI and EPDS, the perinatal and neonatal outcomes such as development and tempoerament of the infants by validated questionnaires AGES and STAGES 6 and 12 months after birth and a follow-up of infants after two years by the Parca-R. questionnaire. In addition the gold MSI will be evaluated in both groups to test the affinity to music as well as the correlation with linguistic development by EEG of the newborns.

Hypothesis: Both interventions lead to a rapid reduction in the psychological and physiological stress of pregnant women. The effects may be more pronounced with live music.

A total of 128 women will be assigned to one of two groups. Taking into account a drop-out rate of 5-10% during the course of the study, the investigators expect to have complete data from 116 women (approximately 58 per group) to evaluate the effectiveness of the intervention.

Based on our previous studies on the reduction of psychological stress and cortisol levels by concert interventions showing significant changes in mean cortisol levels, the effect sizes of the intervention on site are estimated to be moderate: Assuming a moderate effect size (f = 0.25) and a β/α ratio = 4, N = 58 women per group and using 5 repeated measures are needed to detect differences between the two groups.

Due to the fact that the life concerts and workshops had to be prepared by a professional team, the investigators could not perform a randomized controlled trial as orginally intended but hat to form the groups consecutively by recruitment from outpatient units in berlin and environment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 10 gestational weeks onwards not younger than 18 years and not older than 50 years
* no severe medical or mental disease
* capable to understand german or English language

Exclusion Criteria:

* Pregnant women outside the above declared inclusion criteria
* more than 20 gestational weeks at recruitment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women from 12 gestational weeks onwards up to birth.
Enrollment: 200 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Short-term differences before and after musical interventions | Five minutes before and after the workshop or concert starts and ends. In total six concerts and five workshops take place.
  Short-term differences in affection measured immediately before and after all interventions by the PANAS Test (Positive and Negative Affect Schedule). Each time the same six factors are asked in the PANAS. The minimum score is 3 (low affect),the maximum score is 15 (high affect).
Short-term differences before and after musical interventions (Cortisol) | 1. At the second concert (gestational age between 22 and 28 weeks), 2. at the fifth concert (gestational age between 30 and 36 weeks). Not more than three minutes before and after the second and fifth concert.
  Short-term differences in affection measured immediately before and after all interventions by the differences in cortisol level from buccal swabs, measured twice before and after concerts during pregnancy. In the beginning and at the end of the study.

SECONDARY OUTCOMES:
Medium-term outcome measures (PSS) | 1. Gestational age between 12 and 18 weeks, 2. gestational age between 22 and 28 weeks, 3. gestational age between 30 and 36 weeks.
  Changes in maternal mental health throughout pregnancy of validated psychological questionnaires such as PSS (Perceived Stress Scale) from the start of recruitment up to delivery. Minimum score is zero (0) and shows low stress. The maximum score is forty (40) considered as high perceived stress.
Medium-term outcome measures (STAI) | 1. Gestational age between 12 and 18 weeks, 2. gestational age between 22 and 28 weeks, 3. gestational age between 30 and 36 weeks.
  Changes in maternal mental health throughout pregnancy of validated psychological questionnaires such as STAI (State Trait Anxiety Inventory) from the start of recruitment up to delivery. The minimal score result is 10, the maximal score result is 80 for each of the two parts (State and Trait).
Medium-term outcome measures (EPDS) | 1. Gestational age between 12 and 18 weeks, 2. gestational age between 22 and 28 weeks, 3. gestational age between 30 and 36 weeks
  Changes in maternal mental health throughout pregnancy of validated psychological questionnaires such as EPDS (Edinburgh Postnatal Depression Scale) from the start of recruitment up to delivery. The minimal score result is zero (0), thereby 0-9 points signifies low risk of depression. The maximum score result is thirty (30), with more or equal thirteen (13) points demonstrating a high risk for depression. Ten (10) to twelve (12) signifies moderate risk for depression.
Medium-term outcome measures | 1. Gestational age between 12 and 18 weeks, 2. at the end of pregnancy, when women are admitted at the labor room. Since we cannot predict in advance the gestational age at delivery, due to pragmatic reasons, we cannot be more precise.
  Changes in maternal mental health throughout pregnancy by the concentration of cortisol within maternal hair from the start of recruitment up to delivery.
Long-term outcome measures (AGES and STAGES) | 6 and 12 months after birth
  The perinatal and neonatal outcomes as well as follow-up of the infants by AGES and STAGES after 6 and 12 months. The Ages and Stages Questionnaire (ASQ) is a general developmental screening tool that examines developmental challenges at specific ages. Minimum score result is zero (0) and maximum score result is 300. Characterizing the least and the optimal stages of development.
Long-term outcome measures (PARCA-R) | 24 months after birth
  The Parca-R asked at two years after delivery. PARCA-R stands for Parent Report of Children's Abilities-Revised. It is a parent completed questionnaire that can be used to assess children's cognitive and language development at 24 months of age. The minimal value of the PARCA-R score results for a) cognitive and b) language development is zero (0). The maximum of a) is 34 and for b) 50. Thus the minimal value of the total score is zeo (0) and the maximal 84, characterizing the least and the optimal stages of cognitive and verbal development. Within the investigators plan to compare means with ranges to the standards given in the original publication of Johnson et al. (Lancet Child Adolesc Health 2019) and also compare the results of the Live and Digital Group.

OTHER OUTCOMES:
Music performance and development of linguistic skills | 1. Gestational age between 12 and 18 weeks, 2. gestational age between 22 and 28 weeks, 3. gestational age between 30 and 36 weeks
  Goldsmiths musical sophistication index. The minimal score result is 31, representing poor integration of music at home and maximal score result is 266, representing optimal integration of music in every category.
Placental and telomere data from umbilical cord blood a term | Up to 6 months after birth
  EEG (electroencephalogram) of newborns after 3-6 months. Thereby validated questionnaires and, optionally, an EEG device are used, with which the children's brain waves are recorded using non-invasive electrodes that make contact with the skin via a warm gel and are fixed in place with a cap (approx. 5 min resting EEG without acoustic stimulation, approx. 10 min EEG when listening to syllable sequences). The meaning of the tracings with respect of later language development has been established by our group before .
  More specifically, we shall analyze only brain potentials within event-related EEG-tracings, such as mismatch negativity (MMN). Not according to the frequency spectre such as alpha, beta etc. characteristics.
Placental and telomere data from umbilical cord blood a term | Directly after birth
  Telomere length (TL) of the newborns determined at leucocytes in the umbilical blood at birth. Thereby DNA is isolated from whole blood. Leukocyte TL is the most commonly used measure of TL in human epidemiological studies, and it has been postulated that TL dynamics in leukocytes mirror those of the entire hematopoietic stem cell population, the original pool of which is formed early in gestation and serves as the progenitor for cells in all blood lineages.
  Relative TL is measured by quantitative polymerase chain reaction (qPCR), expressed as the ratio of telomere to single-copy gene abundance (T/S ratio), as previously described.
Placental and telomere data from umbilical cord blood a term | Up to 6 months after birth
  Detection of the human placental11β-HSD2 to determine fetal stress during pregnancy.
  Placental 11β-HSD2 protein levels are quantified by Western blotting. The polyclonal sheep anti-human 11β-HSD2 antibody (LOT 318564, The Binding Site Group Ltd, Birmingham, UK) is used and tested beforehand in immunohisto-chemistry on 5 μm paraffin embedded placental sections.
  The blots are incubated overnight with the 11β-HSD2 antibody at a dilution of 1:1000 in 5% skim milk powder and analyzed on the next day. Each blot is repeated at least three times and included an internal control sample that controlled for inter-blotvariability. Protein results are expressed as ratio of 11β- HSD2, to β-Actin (1:80000, LOT GR67149-2, Abcam plc, Cambridge, UK) and expressed as relative optical density units (ROD).

CONTACTS AND LOCATIONS:
Locations (1):
- Clara Angela Foundation Berlin and Foundation of the Berlin Philharmonics, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
We promied to evaluate all data following the german law of data protection and to handle the data anonomously.

REFERENCES:
- [Background] Mannel C, Schaadt G, Illner FK, van der Meer E, Friederici AD. Phonological abilities in literacy-impaired children: Brain potentials reveal deficient phoneme discrimination, but intact prosodic processing. Dev Cogn Neurosci. 2017 Feb;23:14-25. doi: 10.1016/j.dcn.2016.11.007. Epub 2016 Nov 27. PMID 28011436
- [Background] Verner G, Epel E, Lahti-Pulkkinen M, Kajantie E, Buss C, Lin J, Blackburn E, Raikkonen K, Wadhwa PD, Entringer S. Maternal Psychological Resilience During Pregnancy and Newborn Telomere Length: A Prospective Study. Am J Psychiatry. 2021 Feb 1;178(2):183-192. doi: 10.1176/appi.ajp.2020.19101003. Epub 2020 Sep 11. PMID 32911996
- [Background] Faraji J, Soltanpour N, Lotfi H, Moeeini R, Moharreri AR, Roudaki S, Hosseini SA, Olson DM, Abdollahi AA, Soltanpour N, Mohajerani MH, Metz GAS. Lack of Social Support Raises Stress Vulnerability in Rats with a History of Ancestral Stress. Sci Rep. 2017 Jul 13;7(1):5277. doi: 10.1038/s41598-017-05440-8. PMID 28706188
- [Background] Wu Y, Lu YC, Jacobs M, Pradhan S, Kapse K, Zhao L, Niforatos-Andescavage N, Vezina G, du Plessis AJ, Limperopoulos C. Association of Prenatal Maternal Psychological Distress With Fetal Brain Growth, Metabolism, and Cortical Maturation. JAMA Netw Open. 2020 Jan 3;3(1):e1919940. doi: 10.1001/jamanetworkopen.2019.19940. PMID 31995213
- [Background] Olson DM, Bremault-Phillips S, King S, Metz GAS, Montesanti S, Olson JK, Hyde A, Pike A, Hoover T, Linder R, Joggerst B, Watts R. Recent Canadian efforts to develop population-level pregnancy intervention studies to mitigate effects of natural disasters and other tragedies. J Dev Orig Health Dis. 2019 Feb;10(1):108-114. doi: 10.1017/S2040174418001113. Epub 2019 Jan 10. PMID 30626455
- [Background] Entringer S. Prenatal stress exposure and fetal programming of complex phenotypes: interactive effects with multiple risk factors. Neurosci Biobehav Rev. 2020 Oct;117:3-4. doi: 10.1016/j.neubiorev.2020.04.002. Epub 2020 Apr 9. No abstract available. PMID 32278792
- [Background] Braun F, Hardt AK, Ehrlich L, Sloboda DM, Challis JRG, Plagemann A, Henrich W, Braun T. Sex-specific and lasting effects of a single course of antenatal betamethasone treatment on human placental 11beta-HSD2. Placenta. 2018 Sep;69:9-19. doi: 10.1016/j.placenta.2018.07.007. Epub 2018 Jul 11. PMID 30213491
- [Background] Arabin B. Music during pregnancy. Ultrasound Obstet Gynecol. 2002 Nov;20(5):425-30. doi: 10.1046/j.1469-0705.2002.00844.x. No abstract available. PMID 12423477